CLINICAL TRIAL: NCT01734902
Title: Relative Bioavailability Study to Investigate and to Compare Two Different Formulations of Hyoscine Butylbromide, Following Oral Administration in Healthy Male and Female Volunteers (an Open-label, Randomised, Single Dose, Two-way Crossover, Phase I Study)
Brief Title: Relative Bioavailability Study to Investigate and to Compare Two Different Formulations of Hyoscine Butylbromide in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202.846; 2012-003720-20 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-11-23; First posted 2012-11-28 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — Butylscopolammonium Bromide

ARMS (2):
- 1 Hyoscine butylbromide (Experimental): drops, oral administration with 240 mL water
  Interventions: Drug: Hyoscine butylbromide
- 2 Hyoscine butylbromide (Experimental): sugar coated tablets, oral administration with 240 mL water
  Interventions: Drug: Hyoscine butylbromide

INTERVENTIONS:
Drug: Hyoscine butylbromide — sugar coated tablets for oral administration
  Arms: 2 Hyoscine butylbromide
Drug: Hyoscine butylbromide — drops for oral administration
  Arms: 1 Hyoscine butylbromide

SUMMARY:
The objective of the current trial is to establish the bioequivalence of 2 hyoscine butylbromide dose forms following oral administration.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male and female subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2012-12-01 (Actual); Study Completion 2012-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 202.846.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomised, single-dose, open-label, two-way crossover trial in healthy volunteers to investigate and compare the relative bioavailability of two formulations of hyoscine butylbromide administered orally as drops (T: test treatment) or as sugar-coated Buscopan® tablets(R: reference treatment).
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that all subjects met all inclusion/exclusion criteria. Subjects were not to be randomized to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Buscopan® Tablet (R)/Hyoscine Butylbromide Drops (T): Participants administered orally in the morning on Day 1 of period 1 with single dose of 2 sugar-coated tablets of 10 milligram (20 mg) of Buscopan®, followed by 20 mg hyoscine butylbromide drops with dose strength of 2 millilitre (mL) in the morning on Day 1 of period 2, each treatment with 240 mL water. Both treatment periods were separated by a wash-out period of at least 7 days.
- Hyoscine Butylbromide Drops (T)/Buscopan® Tablet (R): Participants administered orally in the morning on Day 1 of period 1 with 20 mg hyoscine butylbromide drops with dose strength of 2 millilitre (mL) orally, followed by single dose of 2 sugar-coated tablets of 10 milligram (20 mg) of Buscopan® in the morning on Day 1 of period 2, each treatment with 240 mL water. Both treatment periods were separated by a wash-out period of at least 7 days.
Period: Overall Study
Arm/Group | Buscopan® Tablet (R)/Hyoscine Butylbromide Drops (T) | Hyoscine Butylbromide Drops (T)/Buscopan® Tablet (R)
Started | 14 | 16
Completed | 14 | 14
Not Completed | 0 | 2
Not completed — Other than listed | 0 | 2

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) :The TS includes all subjects entered in the trial and treated with at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Buscopan® Tablet (R)/Hyoscine Butylbromide Drops (T) | Hyoscine Butylbromide Drops (T)/Buscopan® Tablet (R) | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.1 (8.0) | 37.8 (7.5) | 37.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 5 | 9 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was not captured in this trial.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 14 | 16 | 30
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Measured Concentration of the Hyoscine Butylbromide in Plasma (Cmax)
Description: Cmax, maximum measured concentration of the hyoscine butylbromide in plasma.
Time Frame: Pharmacokinetic samples were collected pre dose at 2 hour (h) and at 0.5, 1, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 6, 8, 10, 14, 24 and 36 h after the drug administration.
Population: Descriptive statistics is based on treated set (TS) and statistical analysis is based on pharmacokinetic (PK) analysis set (PKS). (PKS includes all treated subjects with data for a primary endpoint and without any protocol violation relevant to the statistical evaluation of PK endpoints.)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram/millilitre [pg/mL]
Groups:
- Hyoscine Butylbromide Drops (T): Participants administered orally single dose of 20 mg hyoscine butylbromide drops with dose strength of 2 millilitre (mL) with 240 mL water in the morning on Day 1 of period 1 or period 2.
- Buscopan® Tablet (R): Participants administered orally single dose of 2 sugar-coated tablets of 10 milligram (20 mg) of Buscopan® with 240 mL water in the morning on Day 1 of period 1 or period 2.
Arm/Group | Hyoscine Butylbromide Drops (T) | Buscopan® Tablet (R)
Number analyzed (Participants) | 28 | 28
Picogram/millilitre [pg/mL] | 70.3 (140.0) | 77.1 (167.0)
Statistical Analysis 1: Comparison: Hyoscine Butylbromide Drops (T) vs Buscopan® Tablet (R); Test type: Equivalence — The statistical model, analysis of variance (ANOVA) on the logarithmic scale includes effects: 'sequence', 'subjects within sequences', 'period', and 'treatment'. The effect 'subject within sequences' was considered as random, whereas the other effects were considered as fixed; Adjusted gMean ratio T/R (%) = 86.97, 90% CI 2-sided [74.046 to 102.151], Standard Error of Mean 35.6 — Standard error of the mean is actually intra-individual geometric coefficient variance [%]. Statistical analysis is based on PKS which includes 27 subjects

2. Primary Outcome: Area Under the Concentration-time Curve of the Hyoscine Butylbromide in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: AUC0-tz, area under the concentration-time curve of the hyoscine butylbromide in plasma over the time interval from 0 to the last quantifiable data point
Time Frame: as for outcome 1
Population: Descriptive statistics is based on TS and statistical analysis is based on pharmacokinetic (PK) analysis set (PKS). (PKS includes all treated subjects with data for a primary endpoint and without any protocol violation relevant to the statistical evaluation of PK endpoints.)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hour/millilitre [pg*h/mL]
Arm/Group | Hyoscine Butylbromide Drops (T) | Buscopan® Tablet (R)
Number analyzed (Participants) | 28 | 28
Picogram*hour/millilitre [pg*h/mL] | 564.0 (131.0) | 608.0 (139.0)
Statistical Analysis 1: Comparison: Hyoscine Butylbromide Drops (T) vs Buscopan® Tablet (R); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Adjusted gMean ratio T/R (%) = 89.05, 90% CI 2-sided [77.26 to 102.62], Standard Error of Mean 31.2 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Area Under the Concentration-time Curve of the Hyoscine Butylbromide in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞ )
Description: AUC0-∞, area under the concentration-time curve of the hyoscine butylbromide in plasma over the time interval from 0 extrapolated to infinity
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hour/millilitre [pg*h/mL]
Arm/Group | Hyoscine Butylbromide Drops (T) | Buscopan® Tablet (R)
Number analyzed (Participants) | 28 | 28
Picogram*hour/millilitre [pg*h/mL] | 623.0 (122.0) | 668.0 (125.0)
Statistical Analysis 1: Comparison: Hyoscine Butylbromide Drops (T) vs Buscopan® Tablet (R); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Adjusted gMean ratio T/R [%] = 90.03, 90% CI 2-sided [78.78 to 102.88], Standard Error of Mean 29.3 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From the first dose of trial medication until 7 days after the end of treatment period, upto 9 days.
Arm/Group | Hyoscine Butylbromide Drops (T) | Buscopan® Tablet (R)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 3/30 | 3/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hyoscine Butylbromide Drops (T) (N=30) | Buscopan® Tablet (R) (N=28)
Nausea (Gastrointestinal disorders) | 1 | 2
Headache (Nervous system disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes